CLINICAL TRIAL: NCT07265115
Title: Advanced Preventive Nutritional Supplements Targeting Pathologies in the Preclinical Phase
Brief Title: Preventive Nutritional Supplements for Preclinical Pathologies
Acronym: ALPHANUTRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Edafología y Biología Aplicada del Segura (Other Government)
Collaborators: San Antonio Technologies - San Antonio Catholic University of Murcia (Other)
Responsible Party: Principal Investigator, María-Teresa García-Conesa, Senior Scientist, Centro de Edafología y Biología Aplicada del Segura
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CE042501
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
Keywords: Prediabetes; Natural product; Bioactive compounds; Postprandial glycemia
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: This was a crossover interventional study conducted with 21 volunteers. Volunteers were randomly assigned to receive either the treatment or the placebo twice each. Each participant received both the treatment and the placebo in a sequential manner, with a washout period of two or three days between interventions.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants receive a matching placebo during their assigned period.
  Interventions: Dietary Supplement: Placebo
- Capsules with active ingredients (Experimental): Participants receive the supplement during their assigned period.
  Interventions: Dietary Supplement: Capsules with active ingredients
- Placebo Repetition (Placebo Comparator): This arm was a repetition of the placebo intake
  Interventions: Dietary Supplement: Placebo Repetition
- Capsules with active ingredients Repetition (Experimental): This arm was a repetition of the supplement intake
  Interventions: Dietary Supplement: Capsules with active ingredients Repetition

INTERVENTIONS:
Dietary Supplement: Placebo — Capsules with microcrystalline cellulose 102
  Arms: Placebo
Dietary Supplement: Capsules with active ingredients — Capsules with phloretin rich apple extract, magnesium oxide, cinnamon extract, zinc citrate and chromium picolinate
  Arms: Capsules with active ingredients
Dietary Supplement: Placebo Repetition — Repetition of the placebo (capsules with microcrystalline cellulose 102) intake
  Arms: Placebo Repetition
Dietary Supplement: Capsules with active ingredients Repetition — Repetition of the supplement intake (Capsules with phloretin rich apple extract, magnesium oxide, cinnamon extract, zinc citrate and chromium picolinate)
  Arms: Capsules with active ingredients Repetition

SUMMARY:
The main objective of this intervention study was to evaluate the functionality of a multi-target preparation (rich in dihydrochalcones from apple, chromium picolinate, zinc, magnesium and cinnamon extract) on the glucose response of individuals who show factors associated with prediabetes.

DETAILED DESCRIPTION:
An interventional study was conducted in collaboration with the Catholic University of San Antonio Murcia (UCAM). A total of 21 prediabetic volunteers (fasting blood glucose levels between 100 and 120 mg/dL) who were not taking diabetes medication or antibiotics during the study were recruited.

The participants were invited to an information session to learn more about the study objectives and procedures, and they signed informed consent forms. During this first visit, anthropometric measurements were taken, and a questionnaire was administered to gather information about their diet and physical activity. Each volunteer made four more visits to the UCAM facilities. On each visit, the volunteers ingested either a placebo capsule or the formulated dietary supplement, followed by a standard breakfast consisting of three toasted bread slices and two single-serving packets of strawberry or peach jam (resulting in a total carbohydrate intake of 49.5 g). The volunteers were randomly assigned to receive the placebo or the supplemet and each of them was taken twice. At time 0 and at different times after breakfast intake (15, 30, 45, 60, 75, 90, 105 and 120 min) blood glucose was measured using capillary blood sample obtained by finger prick and a glucometer.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose values between 100 and 120 mg/dL
* To be habitual breakfast consumers

Exclusion Criteria:

* To have diabetes medication during the study
* To have antibiotics during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Incremental Area Under the Curve (iAUC) of blood glucose over 120 minutes | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes and 120 minutes following the consumption of breakfast with each capsule
  Capillary blood glucose was monitored using a glucometer

SECONDARY OUTCOMES:
Peak Blood Glucose Concentration | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes and 120 minutes following the consumption of the breakfast with each capsule
  Maximum post-prandial blood glucose concentration (Cmax) during the 120-minute test period.
Blood Glucose Concentration at different times | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes and 120 minutes following the consumption of the breakfast with each capsule
  Blood glucose concentration at different times post-ingestion
Time to peak concentration for glucose | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes and 120 minutes following the consumption the breakfast with each capsule.
  Time (min) when Cmax of glucose is reached

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Tomás-Barberán, PhD, Principal Investigator — CEBAS-CSIC
Locations (1):
- Universidad Católica de San Antonio (UCAM), Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lira Neto JCG, Damasceno MMC, Ciol MA, de Freitas RWJF, de Araujo MFM, Teixeira CRS, Carvalho GCN, Lisboa KWSC, Marques RLL, Alencar AMPG, Zanetti ML. Efficacy of Cinnamon as an Adjuvant in Reducing the Glycemic Biomarkers of Type 2 Diabetes Mellitus: A Three-Month, Randomized, Triple-Blind, Placebo-Controlled Clinical Trial. J Am Nutr Assoc. 2022 Mar-Apr;41(3):266-274. doi: 10.1080/07315724.2021.1878967. Epub 2021 Feb 19. PMID 33605836
- [Background] Costello RB, Dwyer JT, Saldanha L, Bailey RL, Merkel J, Wambogo E. Do Cinnamon Supplements Have a Role in Glycemic Control in Type 2 Diabetes? A Narrative Review. J Acad Nutr Diet. 2016 Nov;116(11):1794-1802. doi: 10.1016/j.jand.2016.07.015. Epub 2016 Sep 8. PMID 27618575
- [Background] Kostov K. Effects of Magnesium Deficiency on Mechanisms of Insulin Resistance in Type 2 Diabetes: Focusing on the Processes of Insulin Secretion and Signaling. Int J Mol Sci. 2019 Mar 18;20(6):1351. doi: 10.3390/ijms20061351. PMID 30889804
- [Background] Pelczynska M, Moszak M, Bogdanski P. The Role of Magnesium in the Pathogenesis of Metabolic Disorders. Nutrients. 2022 Apr 20;14(9):1714. doi: 10.3390/nu14091714. PMID 35565682
- [Background] Ul Hasnain SZ, Ahmed M, Manzoor R, Amin A, Mudassir J, Jafar Rana S, Abbas K. Anti-inflammatory, antidiabetic and hypolipidemic potential of Cinnamomum verum J. Presi bark coupled with FT-IR and HPLC analysis. Pak J Pharm Sci. 2024 Nov-Dec;37(6):1529-1544. PMID 39923147
- [Background] Zhao F, Pan D, Wang N, Xia H, Zhang H, Wang S, Sun G. Effect of Chromium Supplementation on Blood Glucose and Lipid Levels in Patients with Type 2 Diabetes Mellitus: a Systematic Review and Meta-analysis. Biol Trace Elem Res. 2022 Feb;200(2):516-525. doi: 10.1007/s12011-021-02693-3. Epub 2021 Mar 30. PMID 33783683
- [Background] Georgaki MN, Tsokkou S, Keramas A, Papamitsou T, Karachrysafi S, Kazakis N. Chromium supplementation and type 2 diabetes mellitus: an extensive systematic review. Environ Geochem Health. 2024 Nov 14;46(12):515. doi: 10.1007/s10653-024-02297-5. PMID 39541030
- [Background] Derosa G, Maffioli P, D'Angelo A, Foscaldi V, Piazza R, Mangrella M, Fogacci F, Cicero AFG. Exploring nutraceutical solutions for prediabetes: a narrative review on the effects of banaba and chromium picolinate. Eur Rev Med Pharmacol Sci. 2025 Jun;29(6):324-338. doi: 10.26355/eurrev_202506_37275. PMID 40613623
- [Background] Nakhate KT, Badwaik H, Choudhary R, Sakure K, Agrawal YO, Sharma C, Ojha S, Goyal SN. Therapeutic Potential and Pharmaceutical Development of a Multitargeted Flavonoid Phloretin. Nutrients. 2022 Sep 2;14(17):3638. doi: 10.3390/nu14173638. PMID 36079895